CLINICAL TRIAL: NCT07144670
Title: Evaluating Pericoronary Adipose Tissue Attenuation in Glycometabolic Diseases
Brief Title: Fat Around Heart Arteries as a Measure of Inflammation in Patients With Glycometabolic Disease
Acronym: PCAT-GMD
Status: Active, not recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Katrine Schultz Overgaard, Dr. Med., Odense University Hospital
Other Study IDs: PCAT-GMD
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight; Obesity Type 2 Diabetes Mellitus; Type 2 Diabetes (T2DM); Prediabetes; Inflammation; Adipose Tissue; Adipose Tissue Inflammation
Keywords: inflammation; type 2 diabetes mellitus; diabetes; prediabetes; obesity; pericoronary adipose tissue; PCAT
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2; Prediabetic State; Inflammation; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fasting blood samples included; HbA1c, low-density lipoprotein (LDL), high-density lipoprotein HDL, triglycerides (TG), creatinine, high-sensitivity C-reactive peptide (hs-CRP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obesity (BMI): Categorical: Normal (25-30), overweight (>25-30), obesity 1 (>30-35), obesity 2+ (>35)
- Prediabetes: Categorical: Normal (<39), Prediabtes (39-47 mmol/mol)
- Type 2 Diabetes Mellitus: Categorical: Without diabetes, with diabetes

SUMMARY:
In this study, the objective is to investigate inflammation in the arteries of the heart. A heart CT scan (CCTA) will be used to measure inflammation by assessing the fat tissue surrounding the arteries of the heart. Participants with and without type 2 diabetes who have no heart symptoms have been examined and had a CCTA scan performed.

This study aims to answer the following questions:

• Is inflammation in the surrounding fat tissue of the heart arteries associated with the following glycometabolic conditions: I) Obesity ii) Prediabetes iii) Type 2 diabetes

DETAILED DESCRIPTION:
Background and significance:

Inflammation in the coronary arteries is a key driver of cardiovascular (CV) disease, particularly in individuals with glycometabolic conditions such as obesity and diabetes. However, traditional biomarkers have limited accuracy in detecting coronary inflammation.

Coronary CT angiography (CCTA) allows for the non-invasive measurement of pericoronary adipose tissue (PCAT) attenuation - the fat surrounding coronary arteries. PCAT and the underlying vessels engage in bidirectional communication, and inflammation alters the structure of PCAT, which can be detected by CCTA.

Glycometabolic diseases promote atherosclerosis through endothelial dysfunction and accumulation of inflammatory cells. Obesity and diabetes are both associated with enlarged adipocytes, which may influence PCAT attenuation by lowering its Hounsfield Unit values, potentially masking underlying inflammation. To date, no studies have thoroughly addressed the possibility that PCAT attenuation may be underestimated in this high-risk CV population.

The PCAT-GMD study is a post-hoc analysis of two trials - CARPE-DM (NCT03016910) and DANCAP (NCT04525508) - aiming to evaluate the relationship between PCAT attenuation and the following glycometabolic conditions:

* Obesity (BMI)
* Prediabetes (HbA1c)
* Type 2 diabetes mellitus

Setting and study population:

A single-center cross-sectional, observational study at Odense University Hospital, Svendborg, Denmark. The study enrollment began in March 2016 and ended in July 2019. The study population included 747 cardiovascularly asymptomatic men with and without diabetes.

Examinations:

All participants underwent CCTA.

Additional assessments included:

* Blood pressure and heart rate
* Anthropometrics: height, weight, waist-to-hip ratio
* Blood and urine sampling
* Medical history

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years
* Capable of giving written informed consent

Exclusion Criteria:

* History of CAD
* Symtoms of CAD (angina)
* Any tachyarrhythmias making CCTA impossible
* Estimated glomerular filtration rate (eGFR) under 45 ml/min
* Allergy to iodine contrast
* Critical illness with life expectancy less than 1 year
* Documented heart failure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men
Study Population: CARPE-DM:
  Participants with type 2 diabetes who were cardiac asymptomatic and had no history of CAD. Participants were recruited from the Endocrinology Outpatient Clinic and the Retina Photographhy Clinic at Odense University Hospital, Svendborg, Denmark.
  DANCAP:
  Participants in the age range 65-75 years were recruitted from the large Danish Cardiovascular Screening (DANCAVAS) at Odense University Hospital (OUH), Svendborg Hospital, Denmark. Participants were cardiac asymptomatic and had no history of CAD.
Sampling Method: Non-Probability Sample
Enrollment: 747 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
PCAT Attenuation [Hounsfield Units (HU)] measured by coronary CT angiography | Baseline
  PCAT attenuation [HU] will be assessed for correlation with the following variables:
  * BMI [kg/m²] [Continously, and categorized as normal (ref), overweight, obesity class 1, obesity class 2+].
  * Prediabetes, defined as HbA1c: 39-47 mmol/mol [Categorical: no(ref)/yes].
  * Type 2 diabetes mellitus, defined by WHO criteria [Categorical: no(ref)/yes].

SECONDARY OUTCOMES:
PCAT Attenuation [HU] measured by coronary CT angiography | Baseline
  Analyses will assess whether BMI (kg/m²) mediates the correlation between glycemic status (prediabetes [HbA1c 39-47 mmol/mol, categorical: no/yes] or type 2 diabetes mellitus [WHO criteria], categorical: no/yes] and PCAT attenuation.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, Professor, Principal Investigator — Cardiovascular Research Unit, OUH Svendborg Hospital.
Locations (1):
- Cardiovascular Research Unit, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: No